CLINICAL TRIAL: NCT07228598
Title: Biofilm Formation on Thoracic Drains: Clinical Significance and Association With Antibiotic Resistance
Brief Title: Biofilm on Chest Drains After Thoracic Surgery: Clinical Impact and Antibiotic Resistance
Status: Recruiting | Type: Observational
Sponsor: Caner İşevi, MD (Other)
Responsible Party: Sponsor-Investigator, Caner İşevi, MD, Principal Investigator, Ondokuz Mayıs University
Organization: Ondokuz Mayıs University (Other)
Other Study IDs: B.30.2.ODM.0.20.08/600-660
Record Dates: First submitted 2025-11-13; First posted 2025-11-14 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Biofilms; Thoracic Surgery; Postoperative Infection; Antibiotic Resistance, Bacterial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Biospecimen Retention: Samples Without DNA — Small sections of chest drain tips will be collected for microbiological culture and biofilm analysis. No genetic or DNA-based testing will be performed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group 1 -Short Drain Duration (≤2 Days): Participants whose thoracic chest drains were removed within 2 days after surgery. Drain tip samples from these patients will be analyzed for biofilm formation and microbiological culture.
  Interventions: Other: Chest Drain Tip Sampling
- Group 2 - Moderate Drain Duration (3-4 Days): Participants whose thoracic chest drains remained in place for 3 to 4 days postoperatively. Drain tips will be examined for biofilm presence and bacterial growth patterns.
  Interventions: Other: Chest Drain Tip Sampling
- Group 3 - Long Drain Duration (≥5 Days): Participants with chest drains in place for 5 days or longer. Biofilm formation, bacterial species identification, and antibiotic resistance profiles will be evaluated.
  Interventions: Other: Chest Drain Tip Sampling

INTERVENTIONS:
Other: Chest Drain Tip Sampling — No active intervention; routine chest drain removal followed by microbiological and biofilm analysis of drain tip samples.

SUMMARY:
This prospective observational study aims to investigate the frequency and clinical significance of biofilm formation on thoracic chest drains used after thoracic surgery. Biofilms are structured bacterial communities that adhere to surfaces and can promote infection and antibiotic resistance. In this study, small samples from the tips of chest drains will be collected under sterile conditions at the time of drain removal and analyzed in the microbiology laboratory.

The main objectives are to evaluate the relationship between the duration of chest drain placement and the presence of biofilm, and to identify the antibiotic resistance profiles of microorganisms isolated from these biofilms. Secondary outcomes include the association between biofilm formation, postoperative infections (such as empyema or wound infection), and the length of hospital stay.

This study will be conducted at Ondokuz Mayıs University Faculty of Medicine, Department of Thoracic Surgery, in collaboration with the Department of Microbiology. The findings are expected to contribute to better understanding of optimal drain management and infection prevention strategies after thoracic surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years and older
* Undergoing elective thoracic surgery requiring chest drain placement
* Able and willing to provide written informed consent

Exclusion Criteria:

* Presence of active infection prior to surgery
* Emergency thoracic surgery
* Immunosuppressed patients (e.g., neutropenia, advanced malignancy, organ transplantation)
* Patients receiving systemic antibiotic therapy at the time of drain removal
* Drainage for empyema or pre-existing pleural infection
* Presence of extrathoracic infection focus
* Refusal or inability to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (≥18 years old) who undergo elective thoracic surgery at Ondokuz Mayıs University Faculty of Medicine and require postoperative chest drain placement. Participants are prospectively enrolled and observed until drain removal. Drain tip samples are collected for microbiological and biofilm analysis.
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2025-10-01 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Presence and Intensity of Biofilm Formation on Chest Drain Tips | At the time of chest drain removal (postoperative days 1-7)
  Biofilm formation on the inner surface of chest drain tips will be evaluated using a microplate crystal violet staining method. The optical density (OD) at 492 nm will be measured, and biofilm intensity will be classified according to the Christensen and Chusri scale (non, weak, moderate, strong). The proportion of patients with biofilm-positive drain tips will be recorded and compared across drain duration groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Ondokuz Mayis University Medical Faculty, Department of Thoracic Surgery, Samsun, Samsun, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared because the dataset includes sensitive clinical and microbiological information collected from a single-center study. Data will be used only for the approved research protocol and analyzed in aggregate form to protect participant confidentiality in accordance with institutional and national data protection regulations.